CLINICAL TRIAL: NCT01516749
Title: An Open Label Non-randomized Study Assessing the Efficacy and Tolerability of Fixed-dose Regimen Daily Subcutaneous Anakinra for the Treatment of Moderate to Severe Hidradenitis Suppurativa
Brief Title: Anakinra as a Treatment for Hydradenitis Suppurativa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-08101
Record Dates: First submitted 2011-12-07; First posted 2012-01-25 (Estimated); Results first posted 2014-08-06 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Hidradenitis Suppurativa
Keywords: hidradenitis suppurativa; anakinra
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anakinra (Experimental): All patients in this arm will receive the investigation drug anakinra once daily subcutaneously.
  Interventions: Drug: anakinra

INTERVENTIONS:
Drug: anakinra — Anakinra is supplied in individual pre-filled glass syringes 100mg/0.67mL each. It will be injected subcutaneously once daily for 8 continuous weeks.
  Other Names: Kineret[TM]

SUMMARY:
This is an open-label, proof-of-concept research study to assess the effectiveness of anakinra in the treatment of patients with hidradenitis suppurativa (HS). The planned intervention is to provide about 6 HS patients with anakinra 100mg daily injections to administer subcutaneously for 8 weeks. Then, the study subjects will be followed for a further 8 weeks to monitor for relapse of HS.

ELIGIBILITY:
Inclusion Criteria:

1) Signed informed consent form with Confirmed diagnosis of hidradenitis suppurativa with moderate or severe disease activity

Exclusion Criteria:

1. Use of the following therapies:

   * Etanercept in the 4 weeks prior to the baseline visit (Day 1)
   * Adalimumab in the 8 weeks prior to the baseline visit (Day 1)
   * Infliximab in the 12 weeks prior to the baseline visit (Day 1)
   * Any other investigational biologics in the 8 weeks prior to the baseline visit (Day 1)
   * Leflunomide in the 4 weeks prior to the baseline visit (Day 1) • Thalidomide in the 4 weeks prior to the baseline visit (Day 1)
   * Cyclosporine in the 4 weeks prior to the baseline visit (Day 1)
   * I.V. immunoglobulin (I.V. Ig) in the 8 weeks prior to the baseline visit (Day 1)
   * 6-Mercaptopurine, azathioprine, cyclophosphamide, or chlorambucil in the 12 weeks prior to the baseline visit (Day 1)
   * Colchicine, dapsone, mycophenolate mofetil & systemic antibiotics in the 3 weeks prior to the baseline visit (Day 1)
   * Corticosteroids "20mg/day or >0.4 mg/kg, whichever applies, in the 1 week prior to the baseline visit (Day 1)
2. history of immunocompromise including HIV infection
3. positive Hep B surface antigen -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-10; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kieron S Leslie, M.D., Principal Investigator — University of California, San Francisco - Department of Dermatology
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Background] Revuz JE, Canoui-Poitrine F, Wolkenstein P, Viallette C, Gabison G, Pouget F, Poli F, Faye O, Roujeau JC, Bonnelye G, Grob JJ, Bastuji-Garin S. Prevalence and factors associated with hidradenitis suppurativa: results from two case-control studies. J Am Acad Dermatol. 2008 Oct;59(4):596-601. doi: 10.1016/j.jaad.2008.06.020. PMID 18674845
- [Background] Fitzsimmons JS, Guilbert PR. A family study of hidradenitis suppurativa. J Med Genet. 1985 Oct;22(5):367-73. doi: 10.1136/jmg.22.5.367. PMID 2934550
- [Background] Stojanov S, Kastner DL. Familial autoinflammatory diseases: genetics, pathogenesis and treatment. Curr Opin Rheumatol. 2005 Sep;17(5):586-99. doi: 10.1097/bor.0000174210.78449.6b. PMID 16093838
- [Background] Steinhoff JP, Cilursu A, Falasca GF, Guzman L, Reginato AJ. A study of musculoskeletal manifestations in 12 patients with SAPHO syndrome. J Clin Rheumatol. 2002 Feb;8(1):13-22. doi: 10.1097/00124743-200202000-00005. PMID 17039195
- [Background] Rosi YL, Lowe L, Kang S. Treatment of hidradenitis suppurativa with infliximab in a patient with Crohn's disease. J Dermatolog Treat. 2005 Feb;16(1):58-61. doi: 10.1080/09546630410024547. PMID 15897171
- [Background] Hunger RE, Surovy AM, Hassan AS, Braathen LR, Yawalkar N. Toll-like receptor 2 is highly expressed in lesions of acne inversa and colocalizes with C-type lectin receptor. Br J Dermatol. 2008 Apr;158(4):691-7. doi: 10.1111/j.1365-2133.2007.08425.x. Epub 2008 Jan 30. PMID 18241264
- [Background] Sakai A, Han J, Cato AC, Akira S, Li JD. Glucocorticoids synergize with IL-1beta to induce TLR2 expression via MAP Kinase Phosphatase-1-dependent dual Inhibition of MAPK JNK and p38 in epithelial cells. BMC Mol Biol. 2004 May 4;5:2. doi: 10.1186/1471-2199-5-2. PMID 15125785
- [Background] Leslie KS, Lachmann HJ, Bruning E, McGrath JA, Bybee A, Gallimore JR, Roberts PF, Woo P, Grattan CE, Hawkins PN. Phenotype, genotype, and sustained response to anakinra in 22 patients with autoinflammatory disease associated with CIAS-1/NALP3 mutations. Arch Dermatol. 2006 Dec;142(12):1591-7. doi: 10.1001/archderm.142.12.1591. PMID 17178985
- [Background] Sartorius K, Emtestam L, Jemec GB, Lapins J. Objective scoring of hidradenitis suppurativa reflecting the role of tobacco smoking and obesity. Br J Dermatol. 2009 Oct;161(4):831-9. doi: 10.1111/j.1365-2133.2009.09198.x. Epub 2009 Apr 29. PMID 19438453

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from an academic dermatology practice in San Francisco, CA; informed consent was obtained before study entry.
Pre-assignment Details: 11 patients were screened for inclusion. 6 were eligible and were enrolled.
Period: Active Therapy
Arm/Group | Anakinra
Started | 6
Completed | 5
Not Completed | 1
Not completed — Lost to Follow-up | 1
Period: Follow-up Off Therapy
Arm/Group | Anakinra
Started | 5
Completed | 4
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Eligible per protocol criteria
Arm/Group | Anakinra
Number analyzed (Participants) | 6
Age, Continuous [Mean (Full Range); unit: years] | 37 [27 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 6
Initial modified Sartorius score [Mean (Full Range); unit: units on a scale] — The following are recorded by the dermatologist: (i) anatomical regions involved: axilla, groin, gluteal (left ⁄right) or other region, 3 points per region; (ii) numbers and scores of lesions (nodule 1 point, fistula 6 points) for each region; (iii) longest distance between two relevant lesions (or size of lesion if single) in each region: < 5 cm, 1 point; 5-10 cm, 3 points; > 10 cm, 9 points; and (iv) whether all lesions are separated by normal skin: yes, 0; no (= Hurley III), 9 points. Regional scores are added and summed up to the patient's total score. The upper limit of the scale is open.
  units on a scale | 78.5 [42 to 95]
Initial C-reactive protein [Mean (Standard Deviation); unit: mg/L] — Normal <3.1 mg/L
  mg/L | 30.6 (23.03)

OUTCOME MEASURES:

1. Primary Outcome: Change in Modified Sartorius Score
Description: At each study visit, the same physician (dermatologist) examined patients and recorded the following: (i) anatomical regions involved: axilla, groin, gluteal (left ⁄right) or other region, 3 points per region; (ii) numbers and scores of lesions (nodule 1 point, fistula 6 points) for each region; (iii) longest distance between two relevant lesions (or size of single lesion) in each region: < 5 cm, 1 point; 5-10 cm, 3 points; > 10 cm, 9 points; and (iv) whether all lesions are separated by normal skin: yes, 0; no (= Hurley III), 9 points.
  Regional scores were summed to a total score, ranging from 5 to indefinite. Smaller numbers are better scores and indicate less lesion involvement. Decreases (negative changes) from baseline indicate improvement in disease severity.
Time Frame: Baseline, 8 weeks
Population: The 5 patients who completed 8 weeks of therapy
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Anakinra
Number analyzed (Participants) | 5
units on a scale | -34.8 [-62.05 to -7.56]
Statistical Analysis 1: Comparison: Anakinra; Significance of decrease in modified Sartorius score from Baseline to 8 weeks; Test type: Superiority or Other; p = 0.024, t-test, 2 sided — significance was accepted at p<0.05

2. Secondary Outcome: Change in Quality of Life Assessments
Description: The Physician Global Assessment: The physician assessed disease activity on the visual analog scale ranging from 0mm (absent) to 100mm (worst imaginable).
  The Patient Global Assessment; The patients reported overall (global) disease activity of HS. Patients were asked "What is the overall activity (pain, discharge, odor, and presence of new lesions) of hidradenitis at this visit?" with a scale of 0=no acitivity to 100=maximal activity.
Time Frame: Baseline, 8 weeks
Population: Patients who completed 8 weeks of therapy
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Anakinra
Number analyzed (Participants) | 5
units on a scale
  Physician Global Assessment | -45.8 [-69.5 to -22.1]
  Patient Global Assessment | -35.6 [-61.4 to -9.83]
Statistical Analysis 1: Comparison: Anakinra; Significance of reductions in Physican Global Assessment mean values between baseline and 8 weeks of therapy; Test type: Superiority or Other; p = 0.006, t-test, 2 sided — Significance was accepted at p<0.05
Statistical Analysis 2: Comparison: Anakinra; Significance of reductions in Patient Global Assessment mean values between baseline and 8 weeks of therapy; Test type: Superiority or Other; p = 0.019, t-test, 2 sided — Significance was accepted at p<0.05

3. Secondary Outcome: Change in Dermatology Quality of Life Index (DLQI)
Description: Patient self-administered questionnaire measuring the extent to which disease affects quality of life, range 0-30, with higher score reflecting a larger negative effect of disease on quality of life
Time Frame: Baseline, 8 weeks
Population: Patients who completed 8 weeks of therapy
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Anakinra
Number analyzed (Participants) | 5
units on a scale | -8.4 [-16.57 to -0.23]

4. Secondary Outcome: Change in C-reactive Protein
Description: Change assessed from baseline to end of treatment phase.
Time Frame: Baseline, 8 weeks
Population: Patients who completed 8 weeks of therapy
Measure: Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Anakinra
Number analyzed (Participants) | 5
mg/L | -16.7 [-36.14 to 2.784]

ADVERSE EVENTS:
Time Frame: 16 weeks: 8 weeks of study therapy, followed by an additional 8 weeks of follow-up off therapy
Description: Vital signs and physical examinations were undertaken at every visit. The investigators assessed adverse events throughout the study by direct patient query, observation by study personnel, and spontaneous patient reporting.
Arm/Group | Anakinra
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anakinra (N=6)
Painful injection site (Skin and subcutaneous tissue disorders) | 6 — All patients reported painful injection site reactions, which decreased in severity after a few weeks of treatment.

LIMITATIONS AND CAVEATS:
Limitations of the study include early termination leading to small numbers of subjects analyzed, and lack of control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes